CLINICAL TRIAL: NCT01169935
Title: In Vivo Tracking of Magnetically-labelled Human Mononuclear Cells Using MRI Scanning
Brief Title: Tracking Inflammatory Cells Using Superparamagnetic Particles of Iron Oxide (SPIO) and Magnetic Resonance Imaging (MRI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Translational Medicine Research Collaboration (Other); British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 10/S1102/31
Record Dates: First submitted 2010-07-23; First posted 2010-07-26 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Healthy
Keywords: MRI; SPIO; Healthy Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Administration of Intra-dermal SPIO (Experimental): MRI scanning before and after intra-dermal injection of SPIO.
  Interventions: Drug: Administration of intra-dermal Endorem
- Mantoux, Venesection, Labelled cells (Experimental): Mantoux test then MRI scanning before and after administration of iron-labelled cells obtained by venesection.
  Interventions: Biological: Mantoux test; Biological: Autologous Endorem-labelled mononuclear cells
- Mantoux, Apheresis, Labelled cells (Experimental): Mantoux test then MRI scanning before and after administration of iron-labelled cells obtained by apheresis.
  Interventions: Biological: Mantoux test; Biological: Autologous Endorem-labelled mononuclear cells
- Mantoux, Administration of Endorem (Experimental): Mantoux test then MRI scanning before and after administration of Endorem.
  Interventions: Biological: Mantoux test; Drug: Administration of Endorem
- Mantoux only (Experimental): Mantoux test then serial MRI scanning.
  Interventions: Biological: Mantoux test

INTERVENTIONS:
Drug: Administration of intra-dermal Endorem — single dose, intradermal
  Arms: Administration of Intra-dermal SPIO
Biological: Mantoux test — single dose, intradermal
  Arms: Mantoux only; Mantoux, Administration of Endorem; Mantoux, Apheresis, Labelled cells; Mantoux, Venesection, Labelled cells
Biological: Autologous Endorem-labelled mononuclear cells — single dose, intravenous
  Arms: Mantoux, Apheresis, Labelled cells; Mantoux, Venesection, Labelled cells
Drug: Administration of Endorem — single dose, intravenous
  Arms: Mantoux, Administration of Endorem

SUMMARY:
Treatment of a wide range of diseases using stem cells and other types of cell appears promising. Following administration of cells it is often not clear where exactly the cells have gone and how many of them have reached the target site. This has been one of the challenges of developing these treatment options further. We have developed a method of labelling human cells with a magnetic resonance imaging (MRI) "contrast agent" which contains tiny iron filings. Following intravenous administration it is possible to see where the iron-labelled cells have gone using MRI scanning. We would like to do is to demonstrate that these cells behave normally and migrate to a site of inflammation. We plan to induce an area of inflammation in the forearm of healthy volunteers using the Mantoux test (a test of immunity against tuberculosis) before giving the labelled cells intravenously. After the Mantoux test we will give these volunteers iron-labelled cells and do MRI scans of their forearm to determine whether these cells can be seen accumulating in the target site.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteers age 18 to 65 years
* Previous vaccine for tuberculosis more than 5 years ago

Exclusion Criteria:

* pregnancy / breast feeding
* Contra-indication to MRI scanning
* Inability or refusal to give informed consent
* Renal failure (eGFR <25mL/min) or hepatic dysfunction (Child's B or C)
* HIV/hepatitis B/hepatitis C/HTLV/syphilis
* Active malignant disease
* Anaemia
* Blood dyscrasia
* High risk of allergy to protamine sulphate (fish allergy, infertile men, vasectomy)
* Known history of tuberculosis infection.
* History of prolonged residence (> 6 months) in a region or country with a high prevalence of tuberculosis.
* Previous Mantoux reaction of 15mm of greater.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-07; Primary Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Change in signal intensity in the region of interest on MRI scanning | 0 hours, 24 hours, 48 hours, 3 - 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Jenny M Richards, MBChB MRCS, Principal Investigator — University of Edinburgh
Locations (1):
- University of Edinburgh / Royal Infirmary of Edinburgh, Edinburgh, Scotland, United Kingdom

REFERENCES:
- [Derived] Richards JM, Shaw CA, Lang NN, Williams MC, Semple SI, MacGillivray TJ, Gray C, Crawford JH, Alam SR, Atkinson AP, Forrest EK, Bienek C, Mills NL, Burdess A, Dhaliwal K, Simpson AJ, Wallace WA, Hill AT, Roddie PH, McKillop G, Connolly TA, Feuerstein GZ, Barclay GR, Turner ML, Newby DE. In vivo mononuclear cell tracking using superparamagnetic particles of iron oxide: feasibility and safety in humans. Circ Cardiovasc Imaging. 2012 Jul;5(4):509-17. doi: 10.1161/CIRCIMAGING.112.972596. Epub 2012 Jul 10. PMID 22787016